CLINICAL TRIAL: NCT00651573
Title: Balancing Risk: Red Blood Cell Transfusion Strategies In Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 08-064
Record Dates: First submitted 2008-03-31; First posted 2008-04-03 (Estimated); Results first posted 2019-06-14 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-03

CONDITIONS: Anemia
Keywords: Surgery; Cardiopulmonary bypass; Coronary artery bypass graft; Valve procedure; Hematocrit level; Outcomes
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Blood transfusion triggers of 24% hematocrit value (Active Comparator): Red blood cell transfusion will be given when hematocrit values fall below the assigned group 1 value which is 24%. When the hematocrit value falls to less 24%, a 1 unit RBC transfusion will be administered. Following administration of the 1 unit transfusion a repeat HCT is performed; if the hematocrit value responds to transfusion and is greater than or equal to 24%, no further transfusions will be administered.
  Interventions: Procedure: Blood transfusion at hematocrit value less than 24%
- Blood transfusion triggers of 28% hematocrit value (Active Comparator): Red blood cell transfusion will be given when hematocrit values fall below the assigned group 1 value which is 28%. When the hematocrit value falls to less 28%, a 1 unit RBC transfusion will be administered. Following administration of the 1 unit transfusion a repeat HCT is performed; if the hematocrit value responds to transfusion and is greater than or equal to 28%, no further transfusions will be administered.
  Interventions: Procedure: Blood transfusion at hematocrit value less than 28%

INTERVENTIONS:
Procedure: Blood transfusion at hematocrit value less than 24% — transfusion
  Arms: Blood transfusion triggers of 24% hematocrit value
Procedure: Blood transfusion at hematocrit value less than 28% — transfusion
  Arms: Blood transfusion triggers of 28% hematocrit value

SUMMARY:
The primary purpose of this study is to determine the best blood level to begin transfusing red blood cells in individuals undergoing cardiac surgery.

The secondary aim is to determine the impact of red cell transfusion on health-related quality of life following surgery.

DETAILED DESCRIPTION:
Consecutive consenting patients who meet the inclusion criteria will be randomized to one of 2 transfusion groups based on their HCT value.

Hematocrit Groups:

1. 24%
2. 28%

Red blood cell transfusion will be given only when hematocrit values fall below the assigned group value. When the hematocrit value falls to a value less than the value for the randomized group a 1 unit RBC transfusion will be administered. Following administration of the 1 unit transfusion a repeat HCT is performed; if the hematocrit value responds to transfusion and is greater than or equal to the randomized group no further transfusions will be administered. A measurement of the patient's HCT after each unit of RBC administered is required prior to administering additional units. If a patient's hematocrit is greater than the value for the group which they are randomized, no transfusion of RBC is necessary. Other management decisions are left up to the discretion of the care team. Adherence to the treatment protocol will be required for the patients in the operating room, intensive care unit and postoperatively until discharge from the hospital.

Before surgery, the patient will be asked to respond to a quality-of-life questionnaire. Follow up phone calls will be made by Study personnel at 1 and 3 months after surgery to ask the same questions.

ELIGIBILITY:
Inclusion Criteria:

* All primary and reoperative adult cardiac surgical patients undergoing cardiopulmonary bypass for coronary artery bypass grafting, coronary artery bypass grafting with a valve procedure, isolated valve procedures and ascending aortic repair for aneurysm or dissection procedures.

Exclusion Criteria:

* Age less than 18 years
* Congenital procedures
* Emergencies
* descending thoracic aortic aneurysm repairs
* Left or right ventricular assist devices
* Left ventricular aneurysm resections
* Heart or lung transplantation
* Those unable to receive blood for religious reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 722 (Actual)
Dates: Start 2007-03; Primary Completion 2014-08 (Actual); Study Completion 2019-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel I Sessler, MD, Study Chair — The Cleveland Clinic; Daniel I Sessler, MD, Principal Investigator — The Cleveland Clinic
Locations (2):
- Cleveland Clinic, Cleveland, Ohio, United States
- S.A.L. Hospital and Medical Institute, Ahmedabad, Thaltej,, India

REFERENCES:
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Fergusson DA, Pagano MB, Roubinian NH, Turgeon AF, Valentine S, Trivella M, Doree C, Hebert PC. Transfusion thresholds and other strategies for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2025 Oct 20;10(10):CD002042. doi: 10.1002/14651858.CD002042.pub6. PMID 41114449
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Trivella M, Roubinian N, Fergusson DA, Triulzi D, Doree C, Hebert PC. Transfusion thresholds for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2021 Dec 21;12(12):CD002042. doi: 10.1002/14651858.CD002042.pub5. PMID 34932836

RESULTS

PARTICIPANT FLOW:
Groups:
- Blood Transfusion Triggers of 24% Hematocrit Value: Red blood cell transfusion will be given when hematocrit values fall below the assigned group 1 value which is 24%. When the hematocrit value falls to less 24%, a 1 unit RBC transfusion will be administered. Following administration of the 1 unit transfusion a repeat hematocrit test is performed; if the hematocrit value responds to transfusion and is greater than or equal to 24%, no further transfusions will be administered.
- Blood Transfusion Triggers of 28% Hematocrit Value: Red blood cell transfusion will be given when hematocrit values fall below the assigned group 1 value which is 28%. When the hematocrit value falls to less 28%, a 1 unit RBC transfusion will be administered. Following administration of the 1 unit transfusion a repeat hematocrit test is performed; if the hematocrit value responds to transfusion and is greater than or equal to 28%, no further transfusions will be administered.
Period: Overall Study
Arm/Group | Blood Transfusion Triggers of 24% Hematocrit Value | Blood Transfusion Triggers of 28% Hematocrit Value
Started | 365 | 357
Completed | 363 | 354
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Blood Transfusion Triggers of 24% Hematocrit Value | Blood Transfusion Triggers of 28% Hematocrit Value | Total
Number analyzed (Participants) | 363 | 354 | 717
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (15) | 60 (13) | 60 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 133 | 121 | 254
  Male | 230 | 233 | 463
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 123 | 112 | 235
  India | 240 | 242 | 482
Hematocrit [Median (Inter-Quartile Range); unit: volume percentage of red blood cells] | 37.1 [34.8 to 39.7] | 38.0 [35.0 to 40.2] | 37.6 [35.0 to 40.0]
Serum creatinine [Median (Inter-Quartile Range); unit: mg/dL] | 0.87 [0.75 to 1.05] | 0.87 [0.73 to 1.07] | 0.87 [0.74 to 1.06]

OUTCOME MEASURES:

1. Primary Outcome: A Composite of In-hospital Postoperative Morbidity and Mortality
Description: The composite components were in-hospital mortality, neurologic morbidity (stroke or coma), pulmonary morbidity (pneumonia, pulmonary embolus, or prolonged postoperative ventilation [>24 hours]), renal morbidity (renal failure), infectious morbidity (deep sternal wound infection, septicemia, or sepsis), cardiac arrhythmia (atrial fibrillation, ventricular tachycardia, fibrillation, or asystole), gastrointestinal morbidity, reoperation (for bleeding, tamponade, graft occlusion, valve dysfunction, or noncardiac reasons), and vascular morbidity (aortic or femoral artery dissection or acute limb ischemia).
Time Frame: After surgery until hosptal discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Blood Transfusion Triggers of 24% Hematocrit Value | Blood Transfusion Triggers of 28% Hematocrit Value
Number analyzed (Participants) | 363 | 354
Participants | 59 | 68

2. Secondary Outcome: Length of ICU Stays
Time Frame: After surgery until discharged from ICU
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Blood Transfusion Triggers of 24% Hematocrit Value | Blood Transfusion Triggers of 28% Hematocrit Value
Number analyzed (Participants) | 363 | 354
hours | 67 [56 to 86] | 66 [59 to 72]

3. Secondary Outcome: Length of Hospital Stay
Time Frame: After surgery until hospital discharge
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Blood Transfusion Triggers of 24% Hematocrit Value | Blood Transfusion Triggers of 28% Hematocrit Value
Number analyzed (Participants) | 363 | 354
days | 10 [8 to 11] | 10 [8 to 11]

4. Secondary Outcome: Number of Blood Transfusion
Time Frame: From induction to the end of sugery
Measure: Median (Inter-Quartile Range); unit: times
Arm/Group | Blood Transfusion Triggers of 24% Hematocrit Value | Blood Transfusion Triggers of 28% Hematocrit Value
Number analyzed (Participants) | 363 | 354
times | 1 [0 to 2] | 1 [0 to 3]

5. Secondary Outcome: Prolonged Postoperative Ventilation
Description: On ventilation >24 hours after surgery
Time Frame: After surgeyr until hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Blood Transfusion Triggers of 24% Hematocrit Value | Blood Transfusion Triggers of 28% Hematocrit Value
Number analyzed (Participants) | 363 | 354
Participants | 22 | 18

6. Secondary Outcome: Postoperative Atrial Fibrillation
Time Frame: After surgery until hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Blood Transfusion Triggers of 24% Hematocrit Value | Blood Transfusion Triggers of 28% Hematocrit Value
Number analyzed (Participants) | 363 | 354
Participants | 33 | 45

ADVERSE EVENTS:
Time Frame: After surgery until hospital discharge or 30 days which comes first
Arm/Group | Blood Transfusion Triggers of 24% Hematocrit Value | Blood Transfusion Triggers of 28% Hematocrit Value
All-Cause Mortality (participants affected / at risk) | 0/363 | 0/354
Serious Adverse Events (participants affected / at risk) | 0/363 | 0/354
Other Adverse Events (participants affected / at risk) | 0/363 | 0/354

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes